CLINICAL TRIAL: NCT04368026
Title: Surgical Care in Poland After COVID19 Outbreak - a National Survey Study
Brief Title: SARS-CoV-2 (COVID-19) and Surgery
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Stefura, Reasearch Associate, PhD student at 2nd Department of General Surgery, Principal Investigator, Medical Doctor, Jagiellonian University
Other Study IDs: 1072.6120.103.2020
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Surgical Procedure, Unspecified
MeSH Terms: interventions — Physicians

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Responders currently working in a "COVID-19-dedicated" hospital, which was transformed by Polish Ministry of Health during SARS-CoV-2 pandemic into institution designated only for SARS-CoV-2 patients, including those developing symptoms and quarantined.
  Interventions: Other: No intervention (survey study for medical doctors).
- Group 2: Responders currently working in "non-COVID-19-dedicated" hospital.
  Interventions: Other: No intervention (survey study for medical doctors).

INTERVENTIONS:
Other: No intervention (survey study for medical doctors). — No intervention

SUMMARY:
Importance: During COVID-19 pandemic, it is necessary to collect and analyze data concerning management of hospitals and wards in order to work out solutions for potential future crisis.

Objective: The objective of the study was to investigate how surgical wards in Poland are managing during the COVID-19 pandemic.

Design, Setting and Participants: An anonymous, online survey was designed and published on the official website of The Association of Polish Surgeons. Data was collected between March the 30th and April the 6th of 2020. After data analysis responders were divided into two groups: Group 1 (responders currently working in a "COVID-19-dedicated" hospital) and Group 2 (responders currently working in "non-COVID-19-dedicated" hospital). The study group included Polish surgeons and surgery residents working in surgical departments during pandemic.

DETAILED DESCRIPTION:
Main outcomes and Measures: Descriptive data on perceptions of current status of surgical wards during the pandemic and impact of the pandemic on conducting surgery.

ELIGIBILITY:
Inclusion Criteria:

* The study group included Polish surgeons and surgery residents working in surgical departments during pandemic, who granted an informed consent to participate in the study. .

Exclusion Criteria:

* Retired surgeons, physicians and residents with non-surgical specializations, medical interns, medical students, other health-care professionals were excluded from this study

Min Age: 25 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study group included Polish surgeons and surgery residents working in surgical departments during pandemic.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Descriptive data on perceptions of current status of surgical wards during the pandemic and impact of the pandemic on conducting surgery. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No